CLINICAL TRIAL: NCT07302191
Title: Comparable Reductions in Health Biomarkers Following High-Intensity Interval or Concurrent Training in Obese Postmenopausal Women
Brief Title: High-Intensity Interval or Concurrent Exercise on Oxidative Stress and Inflammation in Obese Women
Acronym: HICONEXOBWO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valladolid (Other)
Collaborators: Sanidad de Castilla y León (Other); Ministerio de Ciencia e Innovación, Spain (Other Government); Fundación General Universidad de Valladolid (Other)
Responsible Party: Principal Investigator, Diego Fernández Lázaro, Professor Doctor, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025.12.11
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Women Veterans; Obese Women; Postmenopausal; Sedentary Lifestlye
Keywords: Concurrent training; High intensity interval training; Postmenopausal women; Obesity; Oxidative stress; Inflammation; Menopause
MeSH Terms: conditions — Obesity; Inflammation | interventions — High-Intensity Interval Training; Control Groups

STUDY DESIGN:
Intervention Model Description: parallel-group randomized controlled
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- high-intensity interval training (HIIT) (Experimental): The HIIT group performed treadmill or overground running/walking intervals consisting of 60 s at 90-95% of maximal heart rate (HRmax), interspersed with 60 s of active recovery at 55-60% HRmax (40) HRmax was estimated individually using the Tanaka et al. equation (41) (HRmax = 208 - 0.7 × age), which has been validated in middle-aged women. Session duration ranged from approximately 25 to 35 min (excluding warm-up and cool-down).
  Interventions: Behavioral: High-Intensity Interval
- Concurrent Training (CONC) (Experimental): The CONC program integrated resistance and aerobic exercise within a single, periodized session designed to elicit both muscular and cardiovascular adaptations.
  Resistance component: Participants performed three sets per exercise targeting major muscle groups (leg press, chest press, seated row, shoulder press, leg curl, and abdominal crunch) with 1 min rest between sets. Training intensity progressed from 55% of one-repetition maximum (1RM) for 10-15 repetitions in week 1 to 75% 1RM for 8-12 repetitions by week 12. To ensure appropriate load progression, 1RM was reassessed every three weeks. Perceived exertion was recorded (Borg 6-20 scale), maintaining RPE 13-15 ("somewhat hard") to confirm compliance with relative intensity.
  Aerobic component: Participants completed 20 min of treadmill running or brisk walking, progressing from 55% HRmax in week 1 to 75% HRmax in week 12, in accordance with the protocol of Kargarfard et al. (44) and consistent with the concurrent training framework
  Interventions: Behavioral: concurrent training
- Control Group (Sham Comparator): Participants assigned to the CG were instructed to maintain their usual daily routines and to refrain from engaging in any structured exercise or new physical activity programs during the 12-week intervention period.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: High-Intensity Interval — HIIT consisted of alternating high- (90-95 % HR_max) and low-intensity (55-60 % HR_max) aerobic bouts
  Arms: high-intensity interval training (HIIT)
Behavioral: concurrent training — combined aerobic and resistance exercises
  Arms: Concurrent Training (CONC)
Behavioral: Control Group — usual daily routines
  Arms: Control Group

SUMMARY:
Introduction: Menopause is associated with body composition change, an increase in the cardio-metabolic risk factor for oxidative stress. Nevertheless, it has been suggested that regular physical training is an effective non-pharmacological intervention to reduce oxidative stress and cardio-metabolic disorders in menopausal individuals. Therefore, the present study was conducted to compare the effects of twelve weeks of high-intensity interval training (HIIT) and concurrent (Conc) and on body composition, cardio-metabolic indices and oxidative stress in sedentary obese postmenopausal women.

Materials and methods: Forty-five menopausal obese women voluntarily participated and were randomly assigned into three groups: a) HIIT (6-12×60s of high intensity training (85-95% HRMax) and then running for 60 seconds with low intensity (55-60% HRMax)), b) concurrent endurance (performed on training with 55-75% HRMax) and strength training (including two sets in eight exercise stations with 55-75% 1RM)) and c) control group. Training programs were done for twelve weeks, 3 times per week. Body composition, cardio-metabolic indices and oxidative stress markers were measured before and after twelve weeks of exercise training program.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least 12 months of amenorrhea.
* Physical abilities with the capacity to exercise safely as determined by a medical evaluation.
* Women in a sedentary state, defined as performing <150 minutes of moderate to vigorous physical activity per week during the previous year.
* BMI >25 and ≤40 kg/ m2

Exclusion Criteria:

* hormone replacement therapy
* smoking.
* diagnosed cardiovascular, renal, or hepatic disease, uncontrolled hypertension, or any musculoskeletal limitation precluding exercise participation

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — sedentary obese postmenopausal women
Enrollment: 58 (Actual)
Dates: Start 2025-09-02 (Actual); Primary Completion 2025-11-20 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Concentration Malondialdehyde (MDA) (nmol/mL) | first day of study and after 80 days of exercise training program (end of study)
  Malondialdehyde (MDA) is a highly reactive compound and a key biomarker for oxidative stress, formed primarily from the breakdown (peroxidation) of polyunsaturated fatty acids in cell membranes, indicating cellular damage
Serum Total Antioxidant Capacity (TAC) | first day of study and after 80 days of exercise training program (end of study)
  Serum Total Antioxidant Capacity (TAC) measures the overall ability of antioxidants in your blood (serum) to neutralize harmful free radicals, reflecting your body's defense against oxidative stress, a key factor in aging and diseases
Concentration Monocyte Chemoattractant Protein-1 (MCP-1) (pg/mL) | first day of study and after 80 days of exercise training program (end of study)
  Monocyte Chemoattractant Protein-1 (MCP-1), also known as CCL2, is a vital CC chemokine that acts as a powerful signal, attracting monocytes, macrophages, and T cells to sites of inflammation, infection, and tissue injury in the body, playing a key role in innate immunity and various inflammatory diseases

SECONDARY OUTCOMES:
Body Mass Index | first day of study and after 80 days of exercise training program (end of study)
  Body Mass Index (BMI) is a simple calculation using your height and weight to estimate body fat
% Body Fat | first day of study and after 80 days of exercise training program (end of study)
  Body fat percentage is the proportion of your total body weight that is fat, not muscle, bone, or water, calculated as (Total Fat Mass / Total Body Mass) x 100
Waist circumference (WC) | first day of study and after 80 days of exercise training program (end of study)
  Waist circumference (WC) is a simple body measurement around your midsection (between the lowest rib and hip bone) used as an indicator of abdominal fat (visceral fat)
hip circumference (HC) | first day of study and after 80 days of exercise training program (end of study)
  Hip circumference (HC) is a key body measurement of the fullest part of your hips and buttocks
waist-hip ratio (WHR) | first day of study and after 80 days of exercise training program (end of study)
  The Waist-to-Hip Ratio (WHR) is a simple measurement dividing your waist circumference by your hip circumference, showing how fat is distributed, especially around your midsection (belly).
total cholesterol (TC) | first day of study and after 80 days of exercise training program (end of study)
  Total Cholesterol (TC) is a blood test measuring all cholesterol in your blood, to assess heart disease risk, with healthy levels generally below 200 mg/dL (or 5.0 mmol/L)
Concentration Triglycerides (TG) (mg/dl) | first day of study and after 80 days of exercise training program (end of study)
  Triglycerides are a common type of fat (lipid) in your blood, serving as the body's main way to store energy from food
Concentration High-Density Lipoprotein Cholesterol (HDL-C) (mg/dl) | first day of study and after 80 days of exercise training program (end of study)
  High-Density Lipoprotein Cholesterol is known as the "good" cholesterol because it helps remove bad cholesterol from your body by transporting it back to the liver for removal
Concentration Low-Density Lipoprotein Cholesterol (LDL-C) (mg/dl) | first day of study and after 80 days of exercise training program (end of study)
  Low-Density Lipoprotein Cholesterol is often called "bad cholesterol" because high levels build up as plaque in your arteries, narrowing them and increasing your risk for heart attacks and strokes, even though high LDL levels usually have no symptoms
Atherogenic Index of Plasma (AIP) | first day of study and after 80 days of exercise training program (end of study)
  he Atherogenic Index of Plasma (AIP) is a key indicator of cardiovascular risk, calculated as the log ratio of triglycerides (TG) to HDL cholesterol (HDL-C) (Log(TG/HDL-C)), reflecting impaired lipid metabolism and inflammation
Serum insulin | first day of study and after 80 days of exercise training program (end of study)
  Serum insulin refers to the amount of the hormone insulin circulating in your blood
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | first day of study and after 80 days of exercise training program (end of study)
  HOMA-IR (Homeostatic Model Assessment of Insulin Resistance) is a calculation that uses your fasting blood glucose and fasting insulin levels to estimate how resistant your body's cells are to insulin.

CONTACTS AND LOCATIONS:
Overall Officials: Diego F Fernández Lázaro, Vice Dean and Professor, Principal Investigator — University of Valladolid
Locations (1):
- Faculty of Health Sciences, University of Valladolid Soria Campus, Soria, Soria 42004, Soria, Spain

IPD SHARING:
Plan to Share IPD: No
It is withheld due to intellectual property rights, to avoid duplication, fear of criticism, time/resource limitations, or to ensure exclusive credit for the initial findings.